CLINICAL TRIAL: NCT05882214
Title: Effect of β-nicotinamide Mononucleotide Intervention on Healthy Young Subjects With Acute Binge Drink: a Double-blinded, Randomized, Crossover Trial
Brief Title: Metabolic Changes Induced by NMN in Healthy Subjects With Acute Binge Drink
Acronym: NMN-MeABD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Li Lab,MD, Professor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Alleviate a hangover with NMN
Record Dates: First submitted 2023-03-16; First posted 2023-05-31 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Binge Drinking; Liver Injury; Nutritional Supplementation; Hepatic Steatosis
Keywords: β-nicotinamide mononucleotide; Acute alcohol intake; Nutritional supplementation; Liver
MeSH Terms: conditions — Binge Drinking; Fatty Liver | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Intervention method using β-nicotinamide mononucleotide
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- maltodextrin group (Placebo Comparator): 4 capsule with 1000mg ''maltodextrin''
  Interventions: Dietary Supplement: Maltodextrin
- β-nicotinamide mononucleotide group (Experimental): 4 capsule with 1000mg ''β-nicotinamide mononucleotide''
  Interventions: Dietary Supplement: β-nicotinamide Mononucleotide

INTERVENTIONS:
Dietary Supplement: β-nicotinamide Mononucleotide — After an 8-hour overnight fast, the participants ingested β-nicotinamide Mononucleotide capsules with a single morning dose of 1000mg. The purity of β-nicotinamide Mononucleotide capsules was no less than 97% according to high-performance liquid chromatography analysis.
  Other Names: NMN
  Arms: β-nicotinamide mononucleotide group
Dietary Supplement: Maltodextrin — After an 8-hour overnight fast, the participants ingested maltodextrin capsules with a single morning dose of 1000mg.
  Arms: maltodextrin group

SUMMARY:
The goal of this double-blinded, randomized, crossover trial is to investigate the effects of NMN supplementation on liver function, liver fat content and lipid metabolism in healthy young subjects with acute binge drink. The main questions it aims to answer are:

1. if NMN administration could accelerate alcohol metabolism and alleviate hangover symptom;
2. if NMN administration could alleviate alcohol-induced liver injury and hepatic steatosis.

DETAILED DESCRIPTION:
The goal of this double-blinded, randomized, crossover trial is to investigate the effects of NMN supplementation on liver function, liver fat content and lipid metabolism in healthy young subjects with acute binge drink. The main questions it aims to answer are:

1. if NMN administration could accelerate alcohol metabolism and alleviate hangover symptom;
2. if NMN administration could alleviate alcohol-induced liver injury and hepatic steatosis.

Participants will be randomized into two groups (n=20), and take 4 NMN capsules (250mg/capsule) or 4 placebo capsules (maltodextrin), respectively. 15 minutes later, they are successively provided with same breakfast and then vodka with a dose of 1g/kg body weight. Venous blood are collected at 0h, 1h, 2h, 3h, 4h, 8h, 12h and 24h from each subject, respectively. In addition, nuclear magnetic resonance imaging (MRI) are taken at 0h, 4h and 24h after alcohol intake. After a 7-day washout period, volunteers are crossed over to another alternative group to receive the corresponding capsules and the test protocol repeats twice.

ELIGIBILITY:
1. Inclusion Criteria:

   a. Sign informed consent
2. Exclusion Criteria:

   1. Neurological disorders
   2. Alcohol allergy
   3. Alcohol addiction
   4. Gastrointestinal diseases
   5. Liver, kidney, cardiovascular or systemic diseases
   6. Antibiotics were administered within 2 weeks prior to the trial
   7. Participants who ate a vegetarian diet
   8. Unable to use a smartphone or computer with Internet access
   9. Participate in another intervention study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Ethanol concentration | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  Ethanol concentration change in mg/dL of each set
Acetaldehyde concentration | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  Acetaldehyde concentration change in mg/dL of each set
Hepatic fibrosis change | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  Research blood hepatic fibrosis include:Hyaluronicacid in ng/mL;Laminin in ng/mL;type Ⅲ in ng/mL;precollagen in ng/mL;type Ⅳ collagen in ng/mL;Fibronect in ng/mL
hepatic function change | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  Research blood hepatic function include:TBIL in μmol/L;Direct bilirubin in μmol/L;Indirect bilirubin in μmol/L;Total bile acid in μmol/L
hepatic injury change | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  Research blood hepatic injury include:Alanine Aminotransferase in U/L;Aspartate Aminotransferase in U/L;Gamma-Glutamyltransferase in U/L;Alpha-Fucosidase in U/L;Alkaline Phosphatase in U/L;cholinesterase in U/L;Lactate Dehydrogenase Enzyme in U/L
Lipid metabolism change | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  Research blood Fat metabolism include:Triglycerides in mmol/L;HDL-Cholesterol in mmol/L;LDL--Cholesterol in mmol/L;Apolipoprotein A in mmol/L;Apolipoprotein B in mmol/L;Lipoprotein(a) in mmol/L
hangover cognition assessment tools after drinking | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  The survey tool consisted of many questions addressing cognition headache, nausea,vomiting,fatigue,concentration,thirst or dehydration,light sensitivity,sleeping difficulty,excessive sweating,anxiety,feelings of depression,trembling or shaking,dizziness,stomachache,and memory loss after drinking

SECONDARY OUTCOMES:
Laboratory markers of inflammation | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  Research blood Inflammatory factor include:Interleukin-2 in pg/ml;Interleukin-4 in pg/ml;Interleukin-6 in pg/ml;Interleukin-8 in pg/ml;Interleukin-10 in pg/ml;Tumor necrosis factor in pg/ml;Interferon gamma in pg/ml;Human IL-1 beta protein in pg/ml;High Sensitivity C-reactive Protein in mg/L
nicotinamide adenine dinucleotide metabolism change | day1-2 and day 8-9 of each 30minutes and 1hour and 2 hours and 3 hours and 4 hours and 5 hours and 6 hours and 12 hours and 24 hours
  NAD+ metabolism will be analysed by performing Liquid Chromatography Mass Spectrometer（LC-MS） on serum
Fecal metabolites | day1-2 and day 8-9 of each set
  Gut microbial communities and their abundant features will be analysed based on shotgun metagenomic sequencing.
Metabolomics profiling | day1-2 and day 8-9 of each set
  Targeted metabonomics are analyzed based on urine and faeces at all visits

CONTACTS AND LOCATIONS:
Overall Officials: Jiaomei Li, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Protect volunteers' personal health data and personal privacy

REFERENCES:
- [Background] Mammen RR, Natinga Mulakal J, Mohanan R, Maliakel B, Illathu Madhavamenon K. Clove Bud Polyphenols Alleviate Alterations in Inflammation and Oxidative Stress Markers Associated with Binge Drinking: A Randomized Double-Blinded Placebo-Controlled Crossover Study. J Med Food. 2018 Nov;21(11):1188-1196. doi: 10.1089/jmf.2017.4177. Epub 2018 Sep 20. PMID 30234415
- [Background] Weissenborn R, Duka T. Acute alcohol effects on cognitive function in social drinkers: their relationship to drinking habits. Psychopharmacology (Berl). 2003 Jan;165(3):306-12. doi: 10.1007/s00213-002-1281-1. Epub 2002 Nov 19. PMID 12439627
- [Background] Kim H, Kim YJ, Jeong HY, Kim JY, Choi EK, Chae SW, Kwon O. A standardized extract of the fruit of Hovenia dulcis alleviated alcohol-induced hangover in healthy subjects with heterozygous ALDH2: A randomized, controlled, crossover trial. J Ethnopharmacol. 2017 Sep 14;209:167-174. doi: 10.1016/j.jep.2017.07.028. Epub 2017 Jul 24. PMID 28750942
- [Background] Lee MH, Kwak JH, Jeon G, Lee JW, Seo JH, Lee HS, Lee JH. Red ginseng relieves the effects of alcohol consumption and hangover symptoms in healthy men: a randomized crossover study. Food Funct. 2014 Mar;5(3):528-34. doi: 10.1039/c3fo60481k. PMID 24458173
- [Background] Torp N, Israelsen M, Nielsen MJ, Astrand CP, Juhl P, Johansen S, Hansen CD, Madsen B, Villesen IF, Leeming DJ, Thiele M, Hansen T, Karsdal M, Krag A. Binge drinking induces an acute burst of markers of hepatic fibrogenesis (PRO-C3). Liver Int. 2022 Jan;42(1):92-101. doi: 10.1111/liv.15120. Epub 2021 Dec 10. PMID 34845832